CLINICAL TRIAL: NCT05476068
Title: Dry Eye Symptoms of University Students Under China's Dynamic COVID-zero Strategy: A Comparison Between the Epidemic and Non-epidemic Areas
Brief Title: Dry Eye Under China's Dynamic COVID-zero Strategy
Status: Completed | Type: Observational
Sponsor: Yifeng Yu (Other)
Responsible Party: Sponsor-Investigator, Yifeng Yu, Deputy chief physician of Ophthalmology center of the Second Affiliated Hospital of Nanchang University, Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Other Study IDs: [2022]NO.(001).
Record Dates: First submitted 2022-07-23; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Dry Eye Symptoms
Keywords: dry eye symptoms; anxiety; depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epidemic area (Nanchang, Nanchang university)
- Non-epidemic area (Kaifeng, Henan university)

SUMMARY:
To compare the prevalence of dry eye symptoms and to investigate the association of the risk factors with the dry eye symptomatology among university students in the epidemic and non-epidemic areas of China under the COVID-zero strategy.

DETAILED DESCRIPTION:
As the COVID-19 outbreak at the end of 2019 spread around the world, the World Health Organization declared it a public health emergency of international concern on 30th January, and a global pandemic on 1st March. In addition to the threat of coronavirus itself, anti-epidemic measures such as wearing masks, maintaining social distance, prohibiting group gathering, blockade, isolation, curfew, closure, working at home, online learning, etc., have also greatly changed people's daily life dynamics. Unlike the previous regional blockade (city-wide) suspension of school and work, China has shifted to dynamic prevention and control in April 2020, and the basic life and activities in the epidemic area are not restricted. This study aims to compare the prevalence of dry eye symptoms and to investigate the association of the risk factors with dry eye symptoms among college students in the epidemic and non-epidemic areas of China under the dynamic COVID-zero strategy.

ELIGIBILITY:
Inclusion criteria:

* College students with age ≥18 years
* No other medication history in recent 2 weeks;
* Have high compliance and are willing to fill in the questionnaire on time

Exclusion criteria:

* routinely using artificial tears and Other eye drops;
* taking any medication that could interfere with the results of the study;
* with any history of eye surgery

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The subjects of the study are students from Nanchang University and Henan University.
Sampling Method: Non-Probability Sample
Enrollment: 1807 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
A score of ocular surface disease index (OSDI)questionnaire | DAY 0
  Ocular surface disease index (OSDI)questionnaire : (1) OSDI: ≤12 (no DED symptoms), 13 ≤ d ≤ 22 (mild DED symptoms), 23 ≤ d ≤ 32 (moderate DED symptoms), and ≥33 (severe DED symptoms).
A score of GAD-7 questionnaire | DAY 0
  GAD-7 questionnaire: (1) 0 < GAD-7 ≤ 4 (normal), 5 ≤ GAD-7 ≤ 9 (mild anxiety), 10 ≤ GAD-7 ≤ 13 (moderate anxiety), 14 ≤ GAD-7 ≤ 18 (moderate and severe anxiety), and 19 ≤ GAD-7 ≤ 21 (severe anxiety).
A score of PHQ-9 questionnaire | DAY 0
  PHQ-9 questionnaire: (1) 0 < PHQ-9 ≤ 4 (normal), 5 ≤ GAD-7 ≤ 9 (mild depression), 10 ≤ GAD-7 ≤ 14 (moderate depression), 15 ≤ GAD-7 ≤ 19 (moderate and severe depression), and 20 ≤ GAD-7 ≤ 27 (severe depression).

SECONDARY OUTCOMES:
A score of UCLA Loneliness Scale questionnaire | DAY 0
  UCLA Loneliness Scale Questionnaire: (1) UCLA < 28 (low loneliness), 28 ≤ UCLA ≤ 33 (generally lower), 33 < UCLA ≤ 39 (intermediate level), 39 < UCLA ≤ 44 (generally higher), and GAD-7 > 44 (highly lonely).
Students' increased use of mobile phones | DAY 0
  Students choose to increase the time of using mobile phones according to options: 0 hours, less than 1 hour, 1-3 hours, 3-5 hours, 5-7 hours, and more than 7 hours
Frequency of student sports | DAY 0
  Students choose the frequency of sports according to the options, which are: less than once a month, 2-3 times a month, 1-2 times a week, 3-5 times a week, and once a day.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No